CLINICAL TRIAL: NCT00545350
Title: Randomized Controlled Trial of Prevention of Fall-related Fractures and Other Injuries by Physical Exercise Among Community Dwelling Elderly Women
Brief Title: Exercise Intervention to Prevent Fall-related Fractures and Other Injuries : The Ossébo Study
Acronym: Ossébo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut national de prevention et d'education pour la sante (Other Government); Partenariats institutions-citoyens pour la recherche et l'innovation, Région Ile de France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AOM06076, K060209; ANR 06BLAN009001,; 047/06-DAS (INPES); 0900342 (Other: PICRI (Région Ile de France))
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2012-05

CONDITIONS: Accidental Falls; Fractures; Fall-related Injuries
Keywords: Prevention; Falls, accidental falls; Fractures; Physical injuries; Women; Elderly; Physical exercise; Balance exercise
MeSH Terms: conditions — Fractures, Bone; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual activity / care
- 2 (Experimental): Physical exercise classes plus home exercises:
  Weekly physical exercise sessions in small groups, led by a qualified and specially trained instructor, and supplemented by simple exercises to do at home. The exercise program will focus on progressive balance retraining but will also include strength/resistance, coordination and flexibility training exercises.
  Interventions: Other: Fall prevention exercise program

INTERVENTIONS:
Other: Fall prevention exercise program — Weekly physical exercise sessions in small groups, led by a qualified and specially trained instructor, and supplemented by simple exercises to do at home.
  The exercise program will focus on progressive balance retraining but will also include strength/resistance, coordination and flexibility training exercises.
  Arms: 2

SUMMARY:
1. Primary objective: to evaluate the effectiveness of a fall prevention exercise program in preventing falls resulting in fractures and other physical traumas.
2. Secondary objectives:

   * to better understand the mechanisms by which physical exercise prevents falls and ensuing injuries (improvement in physical functional abilities, global physical activity level, general physical and psychological wellbeing and self-confidence).
   * to determine the individual factors associated with long-term adherence to the exercise program.

DETAILED DESCRIPTION:
Background : Osteoporotic fractures are a major cause of morbidity and disability in elderly women. Most of these fractures result from a fall. Falls prevention measures largely applicable in the population may contribute to significantly reduce the number of fractures in the population. Recent randomized controlled trials have shown that exercise programs of relatively low intensity, but centered on balance retraining and targeted to subjects at moderate risk, can reduce the risk of falls by 30% in community-dwelling elderly people (Province MA et al 1995 ; Gillepsie LD et al 2003 ; Chang JT et al 2004). But, the effectiveness of exercise in preventing injuries caused by falls, in particular the most serious ones such as those accompanied by fractures, has not been demonstrated. Most previous trials are underpowered to examine the effect of fall prevention exercise programmes on severe injurious falls. Furthermore, there is no consensus about the outcomes of fall related injuries that should be evaluated in controlled trials, and the injurious falls definitions vary substantially across studies. Besides falls leading to fractures and other serious injuries, falls leading to medical care use ought to be considered as well, since their cost for society is high and their burden on the health care system heavy. Falls causing minor injuries are also important, as they may also have serious consequences, such as depression, fear of falling, and activity restriction.

Objectives : To evaluate the effectiveness of exercise in preventing falls resulting in fractures or other physical traumas. Also, to better understand the mechanisms by which physical exercise prevents injurious falls (e.g., improvement in physical functional abilities, global physical activity level, general physical and mental health, and self-confidence), and to determine the individual factors associated with a good long-term adherence to the program.

Method : Randomized controlled trial. Participants will be women aged 75 to 85 years old, living at home, but with impaired physical functional capacity (as assessed by simple functional tests). Women will be recruited using general population lists, such as voter-registration or supplemental health-insurance membership rolls. They will be randomized in 2 groups : one that will receive the intervention, and a control group without it. Each group will include 1000 women followed for 2 years, which will allow to demonstrate a 30% reduction in the frequency of serious falls in the intervention group (if the incidence of serious falls is around 8% per year). Falls and injuries occurrence will be monitored by asking women to return monthly calendar cards where they can mark the date of any falls. A telephone interview will then be realized in case a fall is reported to record the circumstances and consequences of the fall.

Intervention : The intervention will last 2 years and will be implemented in partnership with the association SIEL (Sport, Initiatives, et Loisir) Bleu in 20 study centers located in large and medium-sized cities. It will include weekly exercise sessions in small groups, led by a qualified and specially trained instructor, and supplemented by simple exercises to do at home. The exercise program will focus on progressive balance retraining but will also include strength/resistance, coordination and flexibility training exercises.

Evaluation criteria : The main outcome measure will be the incidence of serious falls defined as " an unexpected event in which the participant comes to rest on the ground, floor, or lower level " and accompanied by a fracture or another serious injury (including head injuries requiring hospitalization, joint dislocations, severe sprains, other non-specified serious joint injuries, and lacerations requiring suturing) (Buchner DM et al 1993). The effectiveness of the intervention on all injurious falls including those leading to more moderate injuries (such as bruises, cuts, abrasions or reduction in physical function for at least 3 days, or if the participant sought medical help (Campbell AJ et al 1997) will also be assessed. Falls associated with an intrinsic major event or an overwhelming hazard (e.g., traffic accident) will be excluded. Intermediate outcome measures, which may help to explain the effect (or absence of effect) of the intervention, will be changes in physical functional capacity (e.g., balance, gait), global physical activity level, feeling of self-efficacy (fear of falling), and general physical and psychological well-being (quality of life). These changes will be evaluated on a sample of participants (160 per group) that will be re-examined at 1 year and 2 years.

Expected results : The group intervention that we propose to assess is relatively simple to implement. It relies on a network of physical exercise instructors already established across France. In case of a demonstrated benefit it could therefore be easily generalized as part of a population-based public health program of fall-related injuries prevention in the elderly. The intervention should enable elderly women to preserve two elements essential to their quality of life as they age, that is, their functional capacity and their independence.

ELIGIBILITY:
Inclusion Criteria:

* women aged 75 years and older,
* living at home but with impaired physical functional capacity (as assessed by simple functional tests: 6-meter walking test and tandem walk test).

Exclusion Criteria:

* serious health problems preventing practice of a physical activity (medical contra-indications),
* already engaged in fall prevention or general group exercise classes.

Ages: 75 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 706 (Actual)
Dates: Start 2007-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of serious fall-related injuries and of all injurious falls including those leading to more moderate injuries | 2 years
  Incidence of serious fall-related injuries (i.e., falls accompanied by fractures, head injuries requiring hospitalization, joint dislocations, severe sprains, other non-specified serious joint injuries, or lacerations requiring suturing), and of all injurious falls including those leading to more moderate injuries (such as bruises, cuts, abrasions or reduction in physical function for at least 3 days, or if the participant sought medical help).

SECONDARY OUTCOMES:
Changes in physical functional capacity, global physical activity level, feeling of self-efficacy (fear of falling), and general physical and psychological well-being (quality of life) at 1 year (mid-intervention) and 2 years (end of intervention) | 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Dargent-Molina, PhD, Principal Investigator — Institut National de la Santé et de la Recherche Médicale, 94800 Villejuif; Bernard Cassou, MD, PhD, Principal Investigator — Université Versailles-Saint Quentin, AP-HP, Hôpital Sainte Périne, 75016, Paris
Locations (20):
- France (20):
  - Hôpital Tenon, Paris, Paris
  - Centre de Recherche Clinique, CHU Amiens Sud, Amiens
  - Centre d'Examen et de Santé (CPAM), Annecy
  - Clinique Les Abondances, Boulogne-Billancourt
  - Centre Hospitalier Universitaire, Caen
  - Hôpital Corentin Celton, Issy-les-Moulineaux
  - Hôpital gériatrique les Bateliers, Lille
  - Centre Régional de Prévention, Lyon
  - Centre de Prévention et de Traitement des Maladies du Vieillissement, CHRU Montpellier, Montpellier
  - Hôpital Bellier (CHU), Nantes
  - Centre d'Examens de Santé (CPAM), Nîmes
  - Hôpital La Collégiale, Paris
  - Centre de Gérontologie Sainte Périne, Paris
  - Observatoire de l'âge, Paris
  - Hôpital Bretonneau, Paris
  - Centre Marnais de Promotion de la Santé, Reims
  - Centre Hospitalier Universitaire Charles Nicolle, Rouen
  - Hôpital de La Charité, Saint-Etienne
  - Hôpital de la Robertsau, Strasbourg
  - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Chang JT, Morton SC, Rubenstein LZ, Mojica WA, Maglione M, Suttorp MJ, Roth EA, Shekelle PG. Interventions for the prevention of falls in older adults: systematic review and meta-analysis of randomised clinical trials. BMJ. 2004 Mar 20;328(7441):680. doi: 10.1136/bmj.328.7441.680. PMID 15031239
- [Background] Buchner DM, Cress ME, de Lateur BJ, Esselman PC, Margherita AJ, Price R, Wagner EH. The effect of strength and endurance training on gait, balance, fall risk, and health services use in community-living older adults. J Gerontol A Biol Sci Med Sci. 1997 Jul;52(4):M218-24. doi: 10.1093/gerona/52a.4.m218. PMID 9224433
- [Background] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Background] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Buchner DM. Falls prevention over 2 years: a randomized controlled trial in women 80 years and older. Age Ageing. 1999 Oct;28(6):513-8. doi: 10.1093/ageing/28.6.513. PMID 10604501
- [Background] Robertson MC, Devlin N, Gardner MM, Campbell AJ. Effectiveness and economic evaluation of a nurse delivered home exercise programme to prevent falls. 1: Randomised controlled trial. BMJ. 2001 Mar 24;322(7288):697-701. doi: 10.1136/bmj.322.7288.697. PMID 11264206
- [Background] Lord SR, Castell S, Corcoran J, Dayhew J, Matters B, Shan A, Williams P. The effect of group exercise on physical functioning and falls in frail older people living in retirement villages: a randomized, controlled trial. J Am Geriatr Soc. 2003 Dec;51(12):1685-92. doi: 10.1046/j.1532-5415.2003.51551.x. PMID 14687345
- [Background] Barnett A, Smith B, Lord SR, Williams M, Baumand A. Community-based group exercise improves balance and reduces falls in at-risk older people: a randomised controlled trial. Age Ageing. 2003 Jul;32(4):407-14. doi: 10.1093/ageing/32.4.407. PMID 12851185
- [Background] Day L, Fildes B, Gordon I, Fitzharris M, Flamer H, Lord S. Randomised factorial trial of falls prevention among older people living in their own homes. BMJ. 2002 Jul 20;325(7356):128. doi: 10.1136/bmj.325.7356.128. PMID 12130606
- [Background] Li F, Harmer P, Fisher KJ, McAuley E, Chaumeton N, Eckstrom E, Wilson NL. Tai Chi and fall reductions in older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2005 Feb;60(2):187-94. doi: 10.1093/gerona/60.2.187. PMID 15814861
- [Background] Gillespie LD, Gillespie WJ, Robertson MC, Lamb SE, Cumming RG, Rowe BH. Interventions for preventing falls in elderly people. Cochrane Database Syst Rev. 2003;(4):CD000340. doi: 10.1002/14651858.CD000340. PMID 14583918
- [Background] Province MA, Hadley EC, Hornbrook MC, Lipsitz LA, Miller JP, Mulrow CD, Ory MG, Sattin RW, Tinetti ME, Wolf SL. The effects of exercise on falls in elderly patients. A preplanned meta-analysis of the FICSIT Trials. Frailty and Injuries: Cooperative Studies of Intervention Techniques. JAMA. 1995 May 3;273(17):1341-7. PMID 7715058
- [Background] Lord SR, Tiedemann A, Chapman K, Munro B, Murray SM, Gerontology M, Ther GR, Sherrington C. The effect of an individualized fall prevention program on fall risk and falls in older people: a randomized, controlled trial. J Am Geriatr Soc. 2005 Aug;53(8):1296-304. doi: 10.1111/j.1532-5415.2005.53425.x. PMID 16078954
- [Background] Tinetti ME, Baker DI, McAvay G, Claus EB, Garrett P, Gottschalk M, Koch ML, Trainor K, Horwitz RI. A multifactorial intervention to reduce the risk of falling among elderly people living in the community. N Engl J Med. 1994 Sep 29;331(13):821-7. doi: 10.1056/NEJM199409293311301. PMID 8078528
- [Background] Robertson MC, Campbell AJ, Gardner MM, Devlin N. Preventing injuries in older people by preventing falls: a meta-analysis of individual-level data. J Am Geriatr Soc. 2002 May;50(5):905-11. doi: 10.1046/j.1532-5415.2002.50218.x. PMID 12028179
- [Background] Kannus P, Sievanen H, Palvanen M, Jarvinen T, Parkkari J. Prevention of falls and consequent injuries in elderly people. Lancet. 2005 Nov 26;366(9500):1885-93. doi: 10.1016/S0140-6736(05)67604-0. PMID 16310556
- [Background] Wolf SL, Barnhart HX, Kutner NG, McNeely E, Coogler C, Xu T. Reducing frailty and falls in older persons: an investigation of Tai Chi and computerized balance training. Atlanta FICSIT Group. Frailty and Injuries: Cooperative Studies of Intervention Techniques. J Am Geriatr Soc. 1996 May;44(5):489-97. doi: 10.1111/j.1532-5415.1996.tb01432.x. PMID 8617895
- [Background] Buchner DM, Hornbrook MC, Kutner NG, Tinetti ME, Ory MG, Mulrow CD, Schechtman KB, Gerety MB, Fiatarone MA, Wolf SL, et al. Development of the common data base for the FICSIT trials. J Am Geriatr Soc. 1993 Mar;41(3):297-308. doi: 10.1111/j.1532-5415.1993.tb06708.x. PMID 8440854
- [Derived] El-Khoury F, Cassou B, Latouche A, Aegerter P, Charles MA, Dargent-Molina P. Effectiveness of two year balance training programme on prevention of fall induced injuries in at risk women aged 75-85 living in community: Ossebo randomised controlled trial. BMJ. 2015 Jul 22;351:h3830. doi: 10.1136/bmj.h3830. PMID 26201510
- [Derived] Castro-Lionard K, Dargent-Molina P, Fermanian C, Gonthier R, Cassou B. Use of calcium supplements, vitamin D supplements and specific osteoporosis drugs among French women aged 75-85 years: patterns of use and associated factors. Drugs Aging. 2013 Dec;30(12):1029-38. doi: 10.1007/s40266-013-0121-9. PMID 24114665